CLINICAL TRIAL: NCT04701268
Title: Pilot Study - Hemiverse Shoulder Prosthesis
Brief Title: Hemiverse Shoulder Prosthesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision Sponsor
Sponsor: 41Hemiverse AG (Industry)
Collaborators: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41H01
Record Dates: First submitted 2020-12-15; First posted 2021-01-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Tears; Hemiarthroplasty
Keywords: total shoulder; failure; salvage; Rotator Cuff Injuries; Rupture; Wounds and Injuries; Shoulder Injuries; Tendon Injuries; hemiverse
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture; Wounds and Injuries; Shoulder Injuries; Tendon Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): Implantation of the Hemiverse Shoulder Prothesis
  Interventions: Other: Device: Hemiverse

INTERVENTIONS:
Other: Device: Hemiverse — Implantation of the hemiverse shoulder prothesis

SUMMARY:
This clinical trial investigates the safety and the preliminary clinical benefit of the hemiverse shoulder prosthesis. Implantation of this newly developed hemi-prosthesis is intended for patients who do not qualify for a regular reverse or hemi-prosthesis due to severe medical conditions, poor bone stock or critical status of the rotator cuff. The expected benefit is, that patients will have a minimally invasive surgical procedure, only addressing the humeral shaft, however with the biomechanical advantage of a total reverse shoulder prosthesis, meaning, that with a minimally invasive surgery a comparable result as with a regular total shoulder prosthesis is accomplished. Patients will be closely monitored within the study protocol for 24 months and thereafter in regular interval as with a normal prosthetic follow-up.

DETAILED DESCRIPTION:
This clinical trial investigates the safety and the preliminary clinical benefit of the hemiverse shoulder prosthesis. Implantation of this newly developed hemi-prosthesis is intended for patients who do not qualify for a regular reverse or hemi-prosthesis due to severe medical conditions, poor bone stock or critical status of the rotator cuff.

To evaluate the clinical condition of the patient a clinical examination including evaluation of the

* Constant-Murley score,
* Subject shoulder value and
* visual analogue scale are performed before inclusion and during the regular follow-ups. To evaluate the bone stock and the musculature a conventional radiological status and a computed tomography of the shoulder will be performed.

Surgical procedure:

A delto-pectoral approach is preferred. The incision starts immediately lateral to the coracoid tip and extends to the insertion of the deltoid on the Humerus. The subscapularis tendon is exposed and detached from the humerus. The humeral head is exposed and dislocated from the joint using an oscillating saw the humeral head is resected. The shaft is prepared to receive a regular humeral stem which is definitely implanted with 0° retroversion. A trial implant is inserted and reduced into the joint. Free mobility of the joint is tested and the stability of the implant documented. According to the trial implants the definite implant is assembled and implanted. After reduction of the implant the subscapularis tendon is reattached to the humerus using transosseous sutures. Regular closure of the incision is performed.

After-care:

Immediately post operatively a anteroposterior radiograph is performed. For the first two post-operative weeks the arm is immobilised in a sling and external rotation is allowed until 0° and flexion until 90° in internal rotation. Thereafter gradual increase of active mobility is allowed until the weeks post operatively, when full load bearing of the arm is allowed. Regular follow-up visits include evaluation of the Constant-Murley score, Subject shoulder value and visual analogue scale. Additionally conventional radiographic status (anteroposterior lateral and axillary view) are performed post-operatively on day 1 or 2, week 6, 4.5 months, 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years
* Cuff failure with associated shoulder destruction which would be suited for hemiarthoplasty
* Shoulder joint destruction in which known alternatives would constitute either a high patient risk or a high functional failure risk.
* Shoulder destruction for which reverse total shoulder replacement would be a high risk for medical reasons (longer operation, more blood loss) or for advanced glenoid bone destruction
* Written informed consent

Exclusion Criteria:

* Systemic contraindication according to internal medical and anesthesiological standards (e.g. Renal disease, Cardiopulmonary Disease, Heart Disease, Medication including Anticoagulation, Poorly controlled diabetes mellitus, Immunosuppressive drugs etc)
* Neuroarthropathy
* Moderate to severe motor axillary nerve dysfunction
* Moderate to severe destruction of deltoid muscle
* Fracture of the scapular spine or displaced fracture of the basis of the acromion
* Fracture of the base of the coracoid
* Destruction of more than superior one third of the humeral shaft
* Chronic inflammatory diseases,which the PI estimates contribute to a higher risk of surgery complications
* Inability to cooperate with postoperative regimen or to understand the trial information
* Impaired judgement

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at day 1 or 2
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at day 7
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at week 6
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at month 4.5
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at month 6
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at month 12
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of a fracture | Assessments will take place after implantation at month 24
  Fracture of the humerus, the scapula and/or the clavicle (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at day 1 or 2
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at day 7
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at week 6
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at month 4.5
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at month 6
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at month 12
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of an infection | Assessments will take place after implantation at month 24
  Infection at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at day 1 or 2
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at day 7
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at week 6
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at month 4.5
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at month 6
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at month 12
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of a hematoma | Assessments will take place after implantation at month 24
  Presence of a hematoma at the implantation site (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at day 1 or 2
  Nerve damage (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at day 7
  Nerve damage (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at week 6
  Nerve damage (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at month 4.5
  Nerve damage (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at month 6
  Nerve damage (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at month 12
  Nerve damage (yes/no).
Adverse Event: Occurence of nerve damage | Assessments will take place after implantation at month 24
  Nerve damage (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at day 1 or 2
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at day 7
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at week 6
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at month 4.5
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at month 6
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at month 12
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of implant dislocation | Assessments will take place after implantation at month 24
  Dislocation of the implant (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at day 1 or 2
  Pulmonary embolism (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at day 7
  Pulmonary embolism (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at week 6
  Pulmonary embolism (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at month 4.5
  Pulmonary embolism (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at month 6
  Pulmonary embolism (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at month 12
  Pulmonary embolism (yes/no).
Adverse Event: Occurence of pulmonary embolism | Assessments will take place after implantation at month 24
  Pulmonary embolism (yes/no).

SECONDARY OUTCOMES:
Change of pain using a visual analogue scale: 0-100, 0=no pain 100=maximal imaginable pain | Assessment will take place at screening and the day before implantation and week 6, month 4.5, month 6, month 12 and month 24
  Highest pain level within last 25 hours will be recorded on a visual analogue scale
Change of active range of motion | Assessment will take place at screening and the day before implantation and week 6, month 4.5, month 6, month 12 and month 24
  Active range of motion of the patient will be measured using a handheld goniometer for active elevation, abduction, external rotation and internal rotation
Change of strength of abduction | Assessment will take place at screening and the day before implantation and week 6, month 4.5, month 6, month 12 and month 24
  isometric strength of abduction will be measured at 90 degrees scapular abduction using a validated device

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Jost, MD, Principal Investigator — Klinik für Orthopädische Chirurgie und Traumatologie des Bewegungsapparates
Locations (1):
- Kantonsspital St. Gallen, Klinik für Orthopädische Chirurgie und Traumatologie des Bewegungsapparates, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No